CLINICAL TRIAL: NCT04670185
Title: Internet-based Parent Training for Parents of Children With Externalising Behavior Problems: A Randomised Controlled Trial
Brief Title: Internet-based Parent Training for Parents of Children With Externalising Behavior Problems
Acronym: BIP-SAMBA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Jens Högström, Associate professor, Karolinska Institutet
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2020-05262
Record Dates: First submitted 2020-12-09; First posted 2020-12-17 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Behavior Problem; Parenting
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet-based parent training (Experimental): Five weeks of therapist-guided online delivered parents training
  Interventions: Behavioral: BIP SAMBA
- Waitlist (No Intervention): Five weeks of waitlist

INTERVENTIONS:
Behavioral: BIP SAMBA — Behavioral parent management training
  Arms: Internet-based parent training

SUMMARY:
The study aims to evaluate the efficacy of a 5-week, therapist-guided, internet-delivered parent management training program (BIP SAMBA) targeting children aged 5 - 11 years with externalising behavior problems. The study is a randomised controlled trial with parents of N=30 children participating. The intervention BIP SAMBA is compared with a waitlist control condition. Participants in the control condition will be crossed over to the active treatment after 5 weeks. The primary outcome measure is the Eyberg Child Behavior Inventory (ECBI) at the post treatment (5 weeks after baseline assessment).

ELIGIBILITY:
Inclusion Criteria:

* Being parent of a child between 5 and 11 years
* This child has externalising behavior problems
* The parent has access to the internet
* The parent speaks and write Swedish

Exclusion Criteria:

* The child has an autism diagnosis
* The child has severe conduct problems
* There is domestic violence occurring within the family
* There alcohol or substance abuse occurring within the family

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
Eyeberg Child Behavior Inventory (ECBI) | Change in conduct problems from baseline (week 0) to post-treatment (week 6)
  Measures externalising behavior problems in children; Min: 0 Max 216; A higher score indicates worse conduct problems.

SECONDARY OUTCOMES:
Strength and Difficulties Questionnaire (SDQ) | Change in mental health issues from baseline (week 0) to post-treatment (week 6)
  Measures conduct problems, emotional problems, ADHD symptoms, peer problems and prosocial behaviours; Min: 0 Max: 40p; A higher score indicate worse mental health problems Screens for behavioral problems, emotional problems, ADHD symptoms, peer problems and pro social behaviours
Alabama Parenting Questionnaire (APQ) | Change in parenting strategies from baseline (week 0) to post-treatment (week 6)
  Measures parenting strategies; Min: 0 Max: 76; A higher score indicates worse parenting strategies
Client Satisfaction Questionnaire (CSQ) | At post-treatment (week 6)
  Measures satisfaction with a treatment that has been received; Min: 0 Max: 24; A higher score indicates better satisfaction with the treatment
Weekly questions about frequency of and impairment from behavior problems | Changes in behavior problems from baseline to week 5
  Participants rate these two questions every week throughout the treatment; Min 0 Max: 9; A higher score indicates worse behavior problems

CONTACTS AND LOCATIONS:
Locations (1):
- BUP CPF, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No